CLINICAL TRIAL: NCT04682665
Title: Biospecimen Collection for:Prebiotic Effect of Eicosapentaenoic Acid Treatment for Colorectal Cancer Liver Metastases
Brief Title: Prebiotic Effect of Eicosapentaenoic Acid Treatment for Colorectal Cancer Liver Metastases
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Massachusetts General Hospital (Other); Massachusetts Institute of Technology (Other); Harvard School of Public Health (HSPH) (Other); University of Bradford (Other)
Responsible Party: Principal Investigator, Mark A Hull, PhD FRCP, Professor of Gastroenterology, University of Leeds
Other Study IDs: 20/YH/0306; 1R01CA243454-01A1 (NIH)
Record Dates: First submitted 2020-12-02; First posted 2020-12-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: Colon Cancer; Liver Metastases; Microbiome
MeSH Terms: conditions — Colonic Neoplasms | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, stool, urine, tumour tissue (colorectal cancer liver metastases).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Experimental: Patients randomized to the experimental arm of the EMT2 trial, receiving Icosapent Ethyl (EPA-EE) according to the EMT2 protocol.
  Interventions: Drug: Icosapent Ethyl Oral Capsule
- Placebo comparator: Patients randomized to the placebo comparator arm of the EMT2 trial, receiving placebo capsules according to the EMT2 protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Icosapent Ethyl Oral Capsule — Soft gelatin capsules containing 1g pure EPA-EE. Administered as 4g per day to be taken as 2 capsules in the morning and 2 capsules in the evening.
  Groups: Experimental
Other: Placebo — Soft gelatin capsules containing light mineral oil. 4 capsules to be taken per day (2 in the morning and 2 in the evening).
  Groups: Placebo comparator

SUMMARY:
A significant proportion of patients who undergo liver surgery to remove bowel cancer that has spread to the liver (metastases) develop disease recurrence and die from the disease. The EMT2 study (NCT03428477) is a clinical trial of the omega-3 fatty acid EPA, investigating whether patients who EPA ethyl ester remain free of disease recurrence for longer than those taking placebo. Recent data suggest that the anti-cancer effect of EPA may result from changes to the microbiota (gut bacteria) which lead to an improved anti-cancer response by the immune system. This study will collect biospecimens (stool, urine, blood, tumour tissue) from participants in the EMT2 trial in order to interrogate the microbiome and immune mechanisms associated with EPA treatment, in relation to participant survival. Insights from this study will identify those most likely to benefit from treatment, leading to more targeted, personalised use of EPA.

DETAILED DESCRIPTION:
Despite advance in the diagnosis and treatment of colorectal cancer (CRC), it remains the second most common cause of cancer-related death in the US and the UK. The majority of deaths from CRC are related to distant metastases, predominantly to the liver.

There are observational and laboratory data supporting the notion that the omega-3 polyunsaturated fatty acid eicosapentaenoic acid (EPA) has anti-CRC activity. These include a phase 2 'window of opportunity' randomised, placebo-controlled trial of EPA provided before surgery for resection of CRC liver metastasis (called the EMT study). A signal that EPA improved progression-free and overall survival after liver surgery provided the rationale for the EMT2 trial, which is a randomised, double-blind placebo-controlled phase 3 trial of the effect of EPA (started before surgery but continued post-operatively) on CRC recurrence and survival after surgery for resectable liver metastases [ClinicalTrials.gov NCT03428477 and EudraCT Number: 2016-000628-24].

The mechanism(s) by which EPA might influence post-operative survival are not well understood. Recent data support the idea that the anti-CRC benefit of EPA may be mediated by modulating the intestinal microbiota and ameliorating tumour-permissive immunosuppressive mechanisms, including inhibition of the activity of regulatory T cells (Tregs) and myeloid-derived suppressor cells (MDSCs), as well as reduced synthesis of inflammatory mediators such as prostaglandin (PG) E2 and chemokine (C-C motif) ligand 2 (CCL2). Mice fed with a high-EPA-containing diet demonstrate 1) increased abundance of gut bacteria, such as Bifidobacterium and Lactobacillus genera that support the host anti-tumour immune response and improve the efficacy of cancer immunotherapy, and 2) decreased abundance of lipopolysaccharide (LPS)-producing bacteria that trigger chronic inflammation and can promote CRC. These data support a hypothesis that a prebiotic effect of EPA abrogates intra-tumoural immunosuppression and ameliorates systemic inflammation to improve survival of CRCLM patients.

EMT2 trial participants are ideally placed to provide biospecimens that can be analysed in order to understand the mechanism(s) of action of EPA given that the laboratory data can eventually be linked to the clinical outcomes from the trial. Biospecimens can be obtained without interference with the EMT2 trial protocol. Stool, urine, and blood samples will be obtained 1) after EMT2 trial randomization, before starting EPA or placebo, 2) just before surgery, and 3) at 6-monthly intervals thereafter, plus liver metastases tumour tissue during surgery. Using these biospecimens, the microbiome and immune pathways altered by EPA will be investigated in relation to participant survival. Mechanistic insights about the anti-CRC activity of EPA from the biospecimen collection project will maximize the knowledge and insights gained from the EMT2 trial and its participants, thereby leading to personalized use of EPA, which will be targeted at those most likely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Only individuals who have already been enrolled in the EMT2 trial are eligible for inclusion in the biospecimen collection study.

Exclusion Criteria:

* There are NO exclusions for entry to the biospecimen collection study if an individual has already been recruited to the EMT2 trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant who has already been enrolled in the EMT2 trial is eligible for inclusion in the biospecimen collection study.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Abundance of individual bacterial taxa in the gut microbiome (eg. Bifidobacterium, Lactobacillus, and Fusobacterium) in stool samples. | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  16S rRNA and metagenomic methods
Microbial gene expression in stool samples | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Bacterial gene expression analysis
Levels of polyunsaturated fatty acids and lipid mediators in stool samples | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Liquid chromatography-mass spectrometric measurement of lipids
Relationship between changes in the gut microbiome induced by EPA and survival of patients | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  16S rRNA and metagenomic methods
Treg cells and myeloid-derived suppressor cells in colorectal cancer liver metastasis tissue | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Immunohistochemistry and flow cytometry for immune cell populations
Levels of expression of immune checkpoint regulators in colorectal cancer liver metastasis tissue | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Immunohistochemistry for CTLA-4, TIGIT, TIM-3, PD-1 in colorectal cancer liver metastasis tissue
Blood levels of chemokines and lipid mediators | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Immunoassay and mass spectrometry of chemokines (plasma CCL2) and lipid metabolites (urinary PGE-M)
Effect of human faecal samples from patients treated with EPA or placebo on tumour burden in gnotobiotic mice with colorectal cancer liver metastasis | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Liver tumour size
Effect of human faecal samples from patients treated with EPA or placebo on anti-tumour immune response in gnotobiotic mice with colorectal cancer liver metastasis | A) Change between baseline (pre-treatment) and before liver surgery. B) Change between baseline (pre-treatment) and 6 months after liver surgery. C) Change between baseline (pre-treatment) and time points up to two years follow up.
  Flow cytometry and immunohistochemistry for immune cell populations and cytokine/chemokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hull, Principal Investigator — University of Leeds
Locations (2):
- United Kingdom (2):
  - St James's University Hospital, Leeds
  - University of Liverpool, Liverpool

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual patient experimental data may be shared depending on experimental outcomes